CLINICAL TRIAL: NCT05630287
Title: A Phase 1, Open-label, Two-part Study to Investigate the Absorption, Metabolism, and Excretion, and the Absolute Bioavailability of [14C]-LOXO-292 in Healthy Male Subjects
Brief Title: A Study of Absorption, Metabolism, Excretion, and Absolute Bioavailability of Carbon-14-Labelled [14C] Selpercatinib (LY3527723) in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17768; J2G-OX-JZJT (Other: Eli Lilly and Company); LOXO-RET-18016 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-11-21; First posted 2022-11-29 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carbon-14-labelled [14C]-Selpercatinib - Part 1 (Experimental): Participants received a single oral dose of 165 milligram (mg) of [14C]-Selpercatinib (containing approximately 40 µCi).
  Interventions: Drug: [14C]-Selpercatinib
- Selpercatinib and [14C]-Selpercatinib - Part 2 (Experimental): Participants received a single oral dose of 160 mg Selpercatinib followed by single dose of <100 µg of [14C]-Selpercatinib (containing approximately 1 µCi) administered intravenously (IV).
  Interventions: Drug: Selpercatinib; Drug: [14C]-Selpercatinib

INTERVENTIONS:
Drug: [14C]-Selpercatinib — Administered as an oral solution
  Other Names: LY3527723; LOXO-292
  Arms: Carbon-14-labelled [14C]-Selpercatinib - Part 1
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292
  Arms: Selpercatinib and [14C]-Selpercatinib - Part 2
Drug: [14C]-Selpercatinib — Administered intravenously
  Other Names: LY3527723; LOXO-292
  Arms: Selpercatinib and [14C]-Selpercatinib - Part 2

SUMMARY:
The main purpose of this study is to compare the amount of selpercatinib that gets into the blood stream and how long it takes the body to get rid of it and also to assess the pharmacokinetics (PK), metabolism, and routes and extent of elimination of selpercatinib in healthy male participants. The study will last up to 59 days (Part 1) or 46 days (Part 2) including screening and 7-day safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study
* Participants will be surgically sterile for at least 90 days prior to Check in or, when sexually active with female partners of childbearing potential, will agree to use effective contraception methods or abstain from sexual intercourse from the time of first dose through 90 days after study drug administration

Exclusion Criteria:

* Participation in any other radiolabeled investigational study drug trial within 12 months prior to Check-in
* Exposure to significant radiation (eg, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to Check-in
* Use or intention to use any medications/products known strong inducers or inhibitors of Cytochrome P450 3A4 enzymes, including St. John's wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LabCorp CRU, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in Part 1 did not participate in Part 2, nor did participants in Part 2 participate in Part 1. Parts 1 and 2 were independent of each other and did not need to be conducted in sequential order.
Groups:
- Selpercatinib and [14C]-Selpercatinib - Part 2: Participants received a single oral dose of 160 mg Selpercatinib followed by a single dose of <100 µg of [14C]-Selpercatinib (containing approximately 1 µCi) administered intravenously (IV).
Period: Overall Study
Arm/Group | Carbon-14-labelled [14C]-Selpercatinib - Part 1 | Selpercatinib and [14C]-Selpercatinib - Part 2
Started | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbon-14-labelled [14C]-Selpercatinib - Part 1 | Selpercatinib and [14C]-Selpercatinib - Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (12.5) | 32 (6.2) | 34 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Selpercatinib in Plasma (Part 1)
Description: PK: AUClast of Selpercatinib in plasma
Time Frame: PK: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- [14C]-Selpercatinib - Part 1: Participants received a single oral dose of 165 milligram (mg) of [14C]-Selpercatinib (containing approximately 40 µCi).
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
hour*nanogram per milliliter (h*ng/mL) | 24100 (20.2)

2. Primary Outcome: PK: AUClast of [14C] Selpercatinib in Plasma and Whole Blood (Part 1) for Total Radioactivity
Description: PK: AUClast of [14C] Selpercatinib in plasma and whole blood
Time Frame: PK: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng equivalents per gram (h*ng Eq/g)
Groups:
- [14C]-Selpercatinib - Part 1: Participants received a single oral dose of 165 mg of [14C]-Selpercatinib (containing approximately 40 µCi).
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
h*ng equivalents per gram (h*ng Eq/g)
  Plasma | 21400 (21.9)
  Whole Blood | 11400 (38.2)

3. Primary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 Extrapolated to Infinity (AUC0-inf) of Selpercatinib in Plasma (Part 1)
Description: PK: AUC0-inf of Selpercatinib in plasma
Time Frame: PK: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
hours*nanogram per milliliter (h*ng/mL) | 24200 (20.2)

4. Primary Outcome: PK: AUC0-inf of [14C] Selpercatinib in Plasma and Whole Blood (Part 1) for Total Radioactivity
Description: PK: AUC0-inf of [14C] Selpercatinib in plasma and whole blood
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng Eq/g
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
h*ng Eq/g
  Plasma | 26900 (25.8)
  Whole Blood | 16700 (32.8)

5. Primary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to Hour 24 (AUC0-24) of Selpercatinib in Plasma (Part 1)
Description: PK: AUC0-24 of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
h*ng/mL | 17100 (17.7)

6. Primary Outcome: PK: (AUC0-24) of [14C] Selpercatinib in Plasma and Whole Blood (Part 1) for Total Radioactivity
Description: PK: AUC0-24 of [14C] Selpercatinib in plasma and whole blood
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng Eq/g
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
h*ng Eq/g
  Plasma | 21400 (21.9)
  Whole Blood | 12600 (23.4)

7. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib in Plasma (Part 1)
Description: PK: Cmax of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
ng/mL | 1890 (22.7)

8. Primary Outcome: PK: Cmax of [14C] Selpercatinib in Plasma and Whole Blood (Part 1) for Total Radioactivity
Description: PK: Cmax of [14C] Selpercatinib in plasma and whole blood
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalents per gram (ng Eq/g)
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
nanogram equivalents per gram (ng Eq/g)
  Plasma | 2240 (24.6)
  Whole Blood | 1260 (25.8)

9. Primary Outcome: PK: Time to Reach Cmax (Tmax) of Selpercatinib in Plasma (Part 1)
Description: PK: Tmax of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
hour (h) | 1.25 [1.00 to 1.50]

10. Primary Outcome: PK: Tmax of [14C] Selpercatinib in Plasma and Whole Blood (Part 1) for Total Radioactivity
Description: PK: Tmax of [14C] Selpercatinib in plasma and whole blood
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: h
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
h
  Plasma | 1.50 [1.00 to 1.50]
  Whole Blood | 1.50 [1.00 to 2.00]

11. Primary Outcome: PK: Apparent First-order Terminal Elimination Half-life (t½) of Selpercatinib in Plasma (Part 1)
Description: PK: t½ of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
h | 36.5 (18.0)

12. Primary Outcome: PK: t½ of [14C] Selpercatinib in Plasma and Whole Blood (Part 1) for Total Radioactivity
Description: PK: t½ of [14C] Selpercatinib in plasma and whole blood
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
h
  Plasma | 12.2 (2.36)
  Whole Blood | 10.5 (2.79)

13. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Selpercatinibin Plasma (Part 1)
Description: PK: CL/F of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
Liter per hour (L/h) | 6.83 (20.2)

14. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Selpercatinib in Plasma (Part 1)
Description: PK: Vz/F of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
Liter (L) | 323 (45.0)

15. Primary Outcome: PK: Plasma Selpercatinib/Total Radioactivity AUC0-24 Ratio (Part 1)
Description: PK: AUC0-24 of Selpercatinib in plasma/AUC0-24 of total radioactivity in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
Ratio | 0.799 (4.4)

16. Primary Outcome: PK: Blood/Plasma Total Radioactivity AUC0-24 Ratio (Part 1)
Description: PK: AUC0-24 of total radioactivity in whole blood/AUC0-24 of total radioactivity in whole blood
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | [14C]-Selpercatinib - Part 1
Number analyzed (Participants) | 6
Ratio | 0.590 (9.0)

17. Primary Outcome: PK: AUClast of Selpercatinib in Plasma (Part 2)
Description: PK: AUClast of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*picogram per mL (h*pg/mL)
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
hour*picogram per mL (h*pg/mL) | 20200 (26.6)

18. Primary Outcome: PK: AUClast of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: AUClast of [14C] Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
h*pg/mL | 1680 (30.0)

19. Primary Outcome: PK: AUC0-inf of Selpercatinib in Plasma (Part 2)
Description: PK: AUC0-inf of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 5
h*pg/mL | 20300 (26.6)

20. Primary Outcome: PK: AUC0-inf of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: AUC0-inf of [14C] Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 5
h*pg/mL | 1720 (33.5)

21. Primary Outcome: PK: Cmax of Selpercatinib in Plasma (Part 2)
Description: PK: Cmax of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
ng/mL | 1550 (28.0)

22. Primary Outcome: PK: Cmax of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: Cmax of [14C] Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
ng/mL | 201 (30.0)

23. Primary Outcome: PK: Tmax of Selpercatinib in Plasma (Part 2)
Description: PK: Tmax of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: h
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
h | 1.92 [1.00 to 1.92]

24. Primary Outcome: PK: Tmax of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: Tmax of [14C] Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: h
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
h | 0.167 [0.167 to 2.10]

25. Primary Outcome: PK: t½ of Selpercatinib in Plasma (Part 2)
Description: PK: t½ of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
h | 31.5 (20.7)

26. Primary Outcome: PK: t½ of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: t½ of [14C] Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 5
h | 16.9 (7.97)

27. Primary Outcome: PK: CL/F of Selpercatinib in Plasma (Part 2)
Description: PK: CL/F of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
L/h | 7.89 (26.6)

28. Primary Outcome: PK: Systemic Clearance (CL) of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: CL of [14C] Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 5
L/h | 5.70 (33.4)

29. Primary Outcome: PK: Vz/F of Selpercatinib in Plasma (Part 2)
Description: PK: Vz/F of Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 6
L | 307 (66.3)

30. Primary Outcome: PK: Volume of Distribution During the Terminal Phase (Vz) of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: Vz of [14C] Selpercatinib in plasma
Time Frame: Pre-dose up to 168 hour post-dose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 5
L | 127 (56.8)

31. Primary Outcome: PK: Volume of Distribution at Steady State (Vss) of [14C] Selpercatinib in Plasma (Part 2)
Description: PK: Vss of [14C] Selpercatinib in plasma
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 5
L | 85.0 (21.0)

32. Primary Outcome: PK: Absolute Bioavailability (F) of Selpercatinib in Plasma (Part 2)
Description: Absolute bioavailability was determined by comparing the plasma exposure of LOXO-292 following oral dosing with the plasma exposure of [14C]-LOXO-292 following IV dosing.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Selpercatinib and [14C]-Selpercatinib - Part 2
Number analyzed (Participants) | 5
Ratio | 0.732 (13.9)

ADVERSE EVENTS:
Time Frame: Part 1: Baseline up to Day 29; Part 2: Baseline up to Day 16
Description: Parts 1 and 2 will consist of all subjects who received at least 1 dose of study drug and have at least 1 post-dose safety assessment.
Groups:
- Carbon-14-labelled [14C]-Selpercatinib: Participants received a single oral dose of 165 milligram (mg) of [14C]-Selpercatinib (containing approximately 40 µCi).
- Selpercatinib and [14C]-Selpercatinib: Participants received a single oral dose of 160 mg Selpercatinib followed by single dose of <100 µg of [14C]-Selpercatinib (containing approximately 1 µCi) administered intravenously (IV).
Arm/Group | Carbon-14-labelled [14C]-Selpercatinib | Selpercatinib and [14C]-Selpercatinib
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbon-14-labelled [14C]-Selpercatinib (N=6) | Selpercatinib and [14C]-Selpercatinib (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT05630287/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT05630287/SAP_001.pdf